CLINICAL TRIAL: NCT03902912
Title: Effect of Prednisolone Treatment on Uterine Natural Killer Cells and Endometrial Angiogenesis in Recurrent Miscarriage Around the Time of Embryo Implantation
Brief Title: Effect of Prednisolone Treatment on Uterine Natural Killer Cells
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.586
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Miscarriage
Keywords: recurrent miscarriage; prednisolone treatment
MeSH Terms: conditions — Abortion, Habitual | interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: The participants will be invited to take prednisolone oral 10 mg/day and attend our outpaitent clinic to be performed endometrial biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prednisolone (Experimental): prednisolone oral 10 mg/day from day one of the subsequent menstrual cycle to day LH plus 7. Women will be then given a tailing off dose of 5 mg/day for 3 days followed by 2 mg/day for 3 days and then 1 mg/day for 3 days.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — prednisolone oral 10 mg/day from day one of the subsequent menstrual cycle to day LH 7 of that cycle. Then, the participants will be given a tailing off dose of 5 mg/day for 3 days followed by 2 mg/day for 3 days and then 1 mg/day for 3 days.

SUMMARY:
This study aims to investigate the role of uNK cells and the association with prednisolone.

DETAILED DESCRIPTION:
Glucocorticoids prednisolone is considered as a potential therapy in women with recurrent miscarriage. However, the evidence for treatment with prednisolone is still inconclusive and the relevant mechanism merits further investigations.

The participants will be invited to take prednisolone oral 10 mg/day and attend our outpaitent clinic to be performed endometrial biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a history of 3 or more consecutive miscarriages
2. Women younger than 40 years old

Exclusion Criteria:

1. Allergy to prednisolone
2. Women who have any uterine anomaly
3. Antiphospholipid syndrome
4. Hydrosalpinx
5. Thrombophilia
6. Abnormal thyroid function tests
7. women with diabetes,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is going to investigate the association between uterine natural killer cells and prednisolone. Therefore, only female will be recruit
Enrollment: 84 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
the number of uNK cells | at the 1 day of endometrial biopsy
  to investigate the association between uNK cells and prednisolone

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided